CLINICAL TRIAL: NCT00749905
Title: A Prospective Randomized Controlled Investigator-blinded Study of Low Fiber Diet for Bowel Preparation for Colon Capsule Examination
Brief Title: Low Fiber Diet for Bowel Preparation for Colon Capsule Examination
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: was not able to recruit enough patients
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Shomron BenHorin, Professor, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SHEBA-08-5217-SBH-CTIL
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Colon Preparation
MeSH Terms: interventions — Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Low fiber diet for 5 days prior to procedure
  Interventions: Other: low fiber diet
- 2 (Active Comparator): regular diet
  Interventions: Other: regular diet

INTERVENTIONS:
Other: low fiber diet — Low fiber diet for 5 days prior to colon capsule
  Arms: 1
Other: regular diet — Regular diet until 1 day before colon capsule
  Arms: 2

SUMMARY:
A prospective randomized controlled investigator-blinded study to compare efficacy of low fiber diet for 5 days versus regular diet, both as adjunct to one day clear liquid diet and standard bowel preparation for colon capsule examination

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and <75
* Colon study indicated for colo-rectal carcinoma screening
* After colonoscopy for any indication failed due to technical causes
* Patients who decline an indicated colonoscopy

Exclusion Criteria:

* Significant heart failure (NYHA grade III-IV)
* Renal failure (Creatinine > 1.2 mg/dl)
* Known or suspected intestinal strictures
* Known or suspected mesenteric adhesions
* History suggestive of bowel obstruction
* Vomiting and/or aspirations
* Symptoms of dysphagia
* Pace-maker or AICD implanted
* Known allergy or intolerance to any of the study drugs
* Pregnancy
* Illicit drug abuse or alcoholism
* Inability to provide an informed consent

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2009-01 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Colon cleanliness | one week from capsule examination

SECONDARY OUTCOMES:
Tolerability of preparations | within 1 day of completing preparation

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel